CLINICAL TRIAL: NCT06243146
Title: Titration of Inspired Oxygen During One-lung Ventilation to Decrease the Incidence of Postoperative Pulmonary Complications: a Randomized Controlled Trial
Brief Title: Titration of Inspired Oxygen to Decrease the Incidence of Postoperative Pulmonary Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Li, Department of Anesthesiology, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SPPH202311011
Record Dates: First submitted 2024-01-28; First posted 2024-02-06 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Unrecognized Condition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Titration (Experimental): During OLV, FiO2 starts at 80%. Titration of inspired oxygen using blood gas analysis and SpO2 monitoring. The titration target is arterial blood gas analysis with PaO2 ≤ 150mmHg and 93% ≤ SpO2 ≤ 97%.
  Interventions: Other: Titration of Inspired Oxygen
- Control (Active Comparator): During OLV, FiO2 starts at 80% and remains until the end of OLV.
  Interventions: Other: Titration of Inspired Oxygen

INTERVENTIONS:
Other: Titration of Inspired Oxygen — Titration of Inspired Oxygen During One-Lung Ventilation

SUMMARY:
Lung cancer is with the highest incidence rate and mortality among people over 60 years old in China. Postoperative pulmonary complications (PPCs) is the most common complication after pneumonectomy, which has a significant impact on the short-term and long-term prognosis of patients, and is even the primary risk factor leading to early postoperative death. High fraction of inspired oxygen (FiO2) is an independent risk factor for PPCs, but it is difficult to achieve oxygenation while avoiding hyperxemia during one lung ventilation (OLV).

We will randomly divide patients who plan to undergo thoracoscopic pulmonary resection into two groups. During OLV, titration will be used to determine the optimal FiO2 for titration group while FiO2 of 80% will be used for mechanical ventilation for control group. The incidence of postoperative PPCs, hypoxia/hyperxemia, severity level of postoperative PPC, postoperative 30 day PPC, increased hospitalization costs, and prolonged hospital stay will be observed in both groups of patients.We will evaluate the effectiveness and safety of titrating inhaled oxygen concentration in lung protection during OLV.

DETAILED DESCRIPTION:
Lung cancer is with the highest incidence rate and mortality among people over 60 years old in China. Postoperative pulmonary complications (PPCs) is the most common complication after pneumonectomy, which has a significant impact on the short-term and long-term prognosis of patients, and is even the primary risk factor leading to early postoperative death. High fraction of inspired oxygen (FiO2) is an independent risk factor for PPCs, but it is difficult to achieve oxygenation while avoiding hyperxemia during one lung ventilation (OLV).Elderly patients with decreased lung function are prone to hypoxemia, which is also a high-risk group for postoperative PPCs induced by hyperxemia, with a dual risk of hypoxia and hyperoxia. Perioperative respiratory management is more challenging. Therefore, it is necessary to explore more suitable oxygen supply methods for patients during OLV.

We will randomly divide patients who plan to undergo thoracoscopic pulmonary resection into two groups. All patients will be intubated with a left bronchial tube using visual laryngoscopy. Fiberoptic bronchoscopy will be used to comfirm the optimal localization of the tube. Lung protective ventilation strategy will be used during ventilation. Before OLV, FiO2 of 100% will be used. During OLV, titration will be used to determine the optimal FiO2 for titration group while FiO2 of 80% will be used for mechanical ventilation for control group. After OLV, FiO2 of 50% will be used. The incidence of postoperative PPCs, hypoxia/hyperxemia, severity level of postoperative PPC, postoperative 30 day PPC, increased hospitalization costs, and prolonged hospital，stay will be compared between 2 groups. The effectiveness and safety of titrating inhaled oxygen concentration during OLV will be elevated.

ELIGIBILITY:
Inclusion Criteria:

* ① General anesthesia with left bronchial tube intubation; ② Age range from 18 to 80 years old; ③ 18 kg/m2 ≤ BMI ≤ 30 kg/m2; ④ ASA grade I to III; ⑤ Individuals willing to participate in research and sign an informed consent form.

Exclusion Criteria:

* ① CT scan indicates preoperative pulmonary infection, atelectasis, and pneumothorax; ② History of respiratory system diseases (COPD, bronchiectasis, pulmonary alveoli, interstitial lung disease, etc.); ③ Previous history of lung surgery; ④ First second forced expiratory volume/estimated value (FEV1%)<60%; ⑤ PaO2<60mmhg (1 mmhg=0.133 kpa) or PaO2/FiO2<300mmhg or SpO2<90% in the suction state; ⑥ History of acute upper respiratory tract infection, acute lung injury, acute respiratory distress syndrome, or respiratory failure within 3 months prior to surgery; ⑦ Combined heart failure (NYHA heart function grading ≥ 3); ⑧ Previous history of stroke and cerebral infarction; ⑨ Severe liver dysfunction (liver failure or Child Pugh score B or C) Chronic renal failure (glomerular filtration rate<30 ml/min) Suffering from mental illness, etc., which is not suitable for the author; æ Individuals who have participated in other clinical trials as subjects within the three months prior to participating in the study The patient refused to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
postoperative pulmonary complications | first 7 days
  postoperative pulmonary complications

CONTACTS AND LOCATIONS:
Overall Officials: Peng Li, MD, Study Chair — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No